CLINICAL TRIAL: NCT01450163
Title: PHASE III, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Pregabalin in Prevention and Reduction of Oxaliplatin-induced Painful Neuropathy
Brief Title: Evaluate The Efficacy and Safety Of Pregabalin In Prevention, Reduction of Oxaliplatin-Induced Painful Neuropathy
Acronym: PreOx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, Dciampi, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PreOx
Record Dates: First submitted 2010-04-26; First posted 2011-10-12 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pain; Neuropathic Pain; Polyneuropathy
Keywords: Neuropathic pain; prevention; prophylaxis; chemotherapy; neuropathy; Oxaliplatin; pregabalin
MeSH Terms: conditions — Pain; Neuralgia; Polyneuropathies | interventions — Pregabalin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin, Oxaliplatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo , Oxaliplatin

INTERVENTIONS:
Drug: Pregabalin, Oxaliplatin — Oxaliplatin will be infused according to the FLOX treatment strategy, as a regular six-month-long adjuvant treatment to colorectal cancer. Pregabalin will be administered P.O. three days before and three days after each of the nine Ox infusions. The dose will be titrated during the first Ox infusion to the highest level tolerated by the patient. The dose used in this first session will be used in the eight following sessions.
  Arms: Pregabalin
Drug: Placebo , Oxaliplatin — Oxaliplatin will be infused according to the FLOX treatment strategy, as a regular six-month-long adjuvant treatment to colorectal cancer. Placebo will be administered P.O. three days before and three days after each of the nine Ox infusions. The dose will be titrated during the first Ox infusion to the highest level tolerated by the patient. The dose used in this first session will be used in the eight following sessions.
  Arms: Placebo

SUMMARY:
Oxaliplatin (Ox) is part of most treatment regimens for colorectal cancer. However, it may induce side effects, such as a specific injury to peripheral nerves called neuropathy. Ox-induced neuropathy is frequently painful. The presence of pain after its administration may hamper the full chemotherapeutic treatment of patients with colorectal cancer receiving this agent. Recently, it has been suggested that the appearance of acute neuropathy after oxaliplatin (Ox) infusion could predict the distal polyneuropathy seen some months after treatment. These two adverse events related to Ox treatment probably share different mechanistic backgrounds. However, recent experimental data suggest that both types of peripheral neuropathies are able to induce central sensitization, a major step to the occurrence of chronic pain. Pregabalin is a molecule used to teat neuropathic pain since it can diminish the peripheral sensitization seen in this painful condition. Recently, it has also been shown that pregabalin can be used to treat neuropathic pain related to Ox treatment. In the present study, we will test the hypothesis that Pregabalin administrated exclusively for three days before and three days after the Ox infusion is able to prevent the occurrence of pain secondary to both the acute and chronic Ox-associated neuropathies. In the classical FLOX chemotherapeutic regimen, Ox is infused in nine sessions during a six-month period. Patients will be followed for a year and nerve conduction tests, quantitative sensory evaluation, pain, quality of life and functional scales will be used to assess the impact of this strategy in the prevention of pain. If this strategy proves to work, this information will have a major impact in the cancer prognosis of patients with colorectal cancer since Ox will be able to administer in its full dose, and will not be limited by neuropathic side effects.

DETAILED DESCRIPTION:
1. OBJECTIVES

1.1. Primary Objectives

The primary objective of this study is to evaluate the efficacy of co-administration of Pregabalin during oxaliplatin infusion in reducing the appearance of both acute and late onset oxaliplatin-induced painful neuropathy in patients with colorectal cancer.

1.2. Secondary Objectives

The secondary objectives of this study are as follows:

* To compare the pain intensity and interference between the two treatment arms
* To compare the safety profile between the two treatment arms
* To compare quality of life between the two treatment arms
* To compare the percentage of patients with neuropathy between the two treatment groups
* To compare the intensity of neuropathy related to oxaliplatin between the two arms
* To compare the small fiber function and positive sensory signs before and after treatment with Pregabalin
* To compare mood (depression and anxiety) before and after treatment with Pregabalin in each treatment arm
* To assess the association between cumulative oxaliplatin dose and time for painful neuropathy and peripheral sensory neuropathy diagnosis, pain intensity, pain interference and small fiber function.

TREATMENT PLAN

2.1 Pregabalin Administration

Treatment will be administered on an outpatient basis. Reported adverse events and potential risks are described in Section 7. Appropriate dose modifications for Pregabalin are described in Section 6. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's oxaliplatin-induced painful neuropathy.

Patients will receive either Pregabalin or placebo three days before and three days following the OX infusion (week 1, 3, and 5 from each of the three cycles, in a total of nine sessions).

The total daily dose of Pregabalin will be flexible in the first dose, and then, a fixed dose will be set for each individual. Before the first Ox dose, patients will start on 75mg bid and will be followed by telephone contact by a research nurse who will instruct them to optimize the dose of Pregabalin every two days according to the magnitude and profile of side effects.

The minimum daily dose to allow for entry in the study is 150mg/day upon the first Ox infusion. Such a "guided" dose escalation will only be performed before the first Ox infusion and will last for four days. Thereafter, the maximum tolerated dose used before the first Ox infusion will be used during the three following days and during the rest of the study. The same protocol will be performed in the placebo group.

After signing the informed consent and agreeing to participate in the protocol, patients will undergo the "guided" Pregabalin dose escalation for four days. Then, they will receive Pregabalin for the three days following the first Ox infusion. Thereafter, they will receive this same Pregabalin dosage for six days during the eight next Ox infusions sessions ie., starting three days before and ending on the third day after each Ox infusion session (from D-3 to D+3)

2.2 Duration of Therapy

In the absence of treatment delays due to adverse event(s), treatment may continue for 3 cycles of FLOX (totalizing nine oxaliplatin infusions) or until one of the following criteria applies:

Intercurrent illness that prevents further administration of treatment,

Unacceptable adverse event(s),

Patient decides to withdraw from the study, or

General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

2.3 FLOX administration

Treatment with fluorouracil plus leucovorin and oxaliplatin (FLOX) 28, 29 will be administered on an outpatient basis.

Patients will receive intravenous (IV) treatment weekly for 6 weeks of each 8-week cycle for three cycles. Chemotherapy with FLOX is to be given for 3 cycles in both treatment arms.

FLOX regimen includes:

* Oxaliplatin will be administered at a dose of 85mg/m2 IV on weeks 1, 3, and 5 of each 8-week cycle for three cycles.
* 5-Fluorouracil (5-FU) will be administered at a dose of 500mg/m2 IV bolus weekly for 6 weeks (on weeks 1, 2, 3, 4, 5, and 6).
* Leucovorin 20 mg/m2 IV will be administered on weeks 1, 2, 3, 4, 5, and 6.

Drugs to be administered before chemotherapy:

Dexamethasone 20 mg IV and Ondansetron 8mg IV will be administered before chemotherapy administration. Dexamethasone will be administered on weeks 1, 3, and 5. Ondansetron will be administered on weeks 1, 2, 3, 4, 5, and 6.

Drugs to be administered after chemotherapy:

Patients will also receive dexamethasone 4 mg P.O. BID for three days and ondansetron 8 mg P.O. each 8 hours (if necessary) after each dose of the Oxaliplatin (on weeks 1, 3, and 5).

2.4 Duration of Follow-up

Patients will be followed for 6 months after removal from study or until death, whichever occurs first. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

2.5 Criteria for study withdraw

After fulfilling all the inclusion criteria and not presenting any exclusion criteria, and having started on the protocol, patients will be removed from it if at least one of the conditions bellow is met:

1. Voluntary consent withdraw by the patients, due to any reason;
2. The patient is considered non compliant to the protocol (ie. more than three absences in regular protocol visits or failure to take Pregabalin for two treatment session with oxaliplatin.

In all cases of removal, the patient data and reason for removal will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed colorectal cancer
* Indication of adjuvant chemotherapy regime including oxaliplatin
* Age ≥ 18 years
* Karnofsky performance status (KPS) ≥ 50
* Normal neurological examination
* Be able to understand study protocol
* Ability to understand and the willingness to sign a written informed consent document.
* The effects of Pregabalin on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* History of exposure to neurotoxic chemotherapy
* Know Concomitant clinical conditions that impair peripheral nerve function,
* Symptoms or signs suggestive of peripheral neuropathy or neuropathic pain.
* Current peripheral neuropathy of NCI-CTCAE, version 3.0 Grade ≥ 1.
* Inadequate organ function, evidenced by the following laboratory results within 1 week prior to randomization:
* Serum creatinine > 2.0 mg/dL
* Positive blood beta HCG test for women, or women breast feeding
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
* History of receiving any investigational treatment within 28 days of randomization
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pregabalin or known hypersensitivity to the study drug.
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy | base line and six months after treatment discontinuation
  Efficacy: the primary endpoint is presence of oxaliplatin-induced painful neuropathy based on Brazilian version of the Douleur Neuropathique 4 Questionnaire (DN4) 1, 2 and intensity of pain based on the numeric pain scale (11-points) of the Brief Pain Inventory.

SECONDARY OUTCOMES:
Safety | base line and six months after treatment discontinuation
  1.Safety:Incidence and severity of adverse (AEs) and serious adverse events (SAEs); 2.Quality of life/Patient report outcomes, European Organization for Research and Treatment of Cancer Quality of Life Questionnaire(EORTC-QLQ-C30);3.Large and small fiber nerve function(Nerve conduction tests -NCT);4.Pain intensity and interference(Brief Pain Inventory-BPI);5.Depression and Anxiety (Hospital Anxiety and Depression Scale-HADS);6.Medication use(Medication Quantification Scale-MQS);7.Oxaliplatin related Neuropathy,Common Toxicity Criteria and the Total Neuropathy Scale (TNS).
Quality of Life | base line and six months after treatment discontinuation
  This study will use the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire- Core (EORTC-QLQ-C30) version 3.0. The EORTC-QLQ-C30 provides a QoL score on physical, role, emotional, cognitive and social functioning; a global health status; and symptom scales (pain, constipation, fatigue, and nausea and vomiting).
Presence of large and small fiber injury | base line and six months after treatment discontinuation
  Peripheral nerve conduction will be assessed by the Nerve conduction tests (NCT) in the upper and lower limbs (ulnar, radial, sural, and peroneal nerves) and samll fiber function will be assessed y a quantitative sensory system protocol 7. Evaluations will take place before, at six and 12 months after study start.
Cancer treatment efficacy | six months after treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C de Andrade, MD, PhD, Principal Investigator — ICESP, Departamento de Neurologia do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo ICESP, São Paulo, Brazil

REFERENCES:
- [Derived] de Andrade DC, Jacobsen Teixeira M, Galhardoni R, Ferreira KSL, Braz Mileno P, Scisci N, Zandonai A, Teixeira WGJ, Saragiotto DF, Silva V, Raicher I, Cury RG, Macarenco R, Otto Heise C, Wilson Iervolino Brotto M, Andrade de Mello A, Zini Megale M, Henrique Curti Dourado L, Mendes Bahia L, Lilian Rodrigues A, Parravano D, Tizue Fukushima J, Lefaucheur JP, Bouhassira D, Sobroza E, Riechelmann RP, Hoff PM; PreOx Workgroup; Valerio da Silva F, Chile T, Dale CS, Nebuloni D, Senna L, Brentani H, Pagano RL, de Souza AM. Pregabalin for the Prevention of Oxaliplatin-Induced Painful Neuropathy: A Randomized, Double-Blind Trial. Oncologist. 2017 Oct;22(10):1154-e105. doi: 10.1634/theoncologist.2017-0235. Epub 2017 Jun 26. PMID 28652279